CLINICAL TRIAL: NCT03754751
Title: Modified Enhanced Recovery Program in Patients With Acute Cholecystitis Undergoing Laparoscopic Cholecystectomy: Prospective Randomized Trial
Brief Title: Enhanced Recovery in Laparoscopic Cholecystectomy
Acronym: ERLAC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pirogov Russian National Research Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ERLAC
Record Dates: First submitted 2018-11-21; First posted 2018-11-27 (Actual); Last update posted 2021-01-15 (Actual); Status verified 2019-11

CONDITIONS: Acute Cholecystitis; Gangrenous Cholecystitis
Keywords: enhanced recovery; intraperitoneal anesthesia; low pressure pneumoperitoneum; cholecystitis; in-hospital stay; laparoscopic cholecystectomy
MeSH Terms: conditions — Cholecystitis, Acute; Cholecystitis | interventions — Cholecystectomy, Laparoscopic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Modified ERAS program group (Experimental): Laparoscopic cholecystectomy with the implementation of modified ERAS program
  Interventions: Procedure: Laparoscopic cholecystectomy with the implementation of modified ERAS program
- Conventional care group (Active Comparator): Laparoscopic cholecystectomy with standard perioperative treatment
  Interventions: Procedure: Laparoscopic cholecystectomy with standard perioperative treatment

INTERVENTIONS:
Procedure: Laparoscopic cholecystectomy with the implementation of modified ERAS program — Preoperative Crystalloid isotonic solutions and antibiotic prophylaxis 30 min prior to surgery.
  1) Patient informing and brochure
  Surgery Cholecystectomy using monopolar by experienced surgeons under general anesthesia
  1. Low-pressure pneumoperitoneum (8-9 mmHg)
  2. Trocar wound and intraabdominal anesthesia with 0.25% ropivacaine
  3. PONV prophylaxis in patients of risk
  Postoperative care
  1. Early mobilization (2 h after surgery)
  2. Early fluid intake (2 h after surgery)
  3. Early liquid food (6 h after surgery) Antibiotics for 3-5 d for patients with complicated cholecystitis (TG13 2). The postoperative pain level evaluation in rest by VAS in 0 h (immediately after awakening), 6 h and 24 h postop. The postoperative analgesic modality "on demand": Ketorolac 30 mg for patients with VAS pain level ≥ 5 cm. Antiemetics in dyspepsia. No iv infusions postoperatively. Intestinal peristalsis evaluation by auscultation every 2 h after surgery
  Arms: Modified ERAS program group
Procedure: Laparoscopic cholecystectomy with standard perioperative treatment — Preoperative Crystalloid isotonic solutions and antibiotic prophylaxis 30 min prior to surgery.
  1) Patient oral informing. No brochure
  Surgery Cholecystectomy using monopolar by experienced surgeons under general anesthesia
  1. Standard CO2 pressure (12-14 mmHg)
  2. No additional anesthesia
  Postoperative care
  1. Mobilization in 4-6 h after surgery
  2. Fluid intake in 6 hours
  3. Liquid food intake in 12 hours Antibiotics for 3-5 d for patients with complicated cholecystitis (TG13 2). The postoperative pain level evaluation in rest by VAS in 0 h (immediately after awakening), 6 h and 24 h postop. The postoperative analgesic modality "on demand": Ketorolac 30 mg for patients with VAS pain level ≥ 5 cm. Antiemetics in dyspepsia. No iv infusions postoperatively. Intestinal peristalsis evaluation by auscultation every 2 h after surgery
  Arms: Conventional care group

SUMMARY:
The study assesses the impact of the modified enhanced recovery protocol on the results of surgical treatment of patients with acute cholecystitis.

DETAILED DESCRIPTION:
Laparoscopic cholecystectomy (LC) is the most common surgical procedures in the world. Elective LC is commonly performed as one-day surgery, while in an emergency setting of acute cholecystitis the in-hospital stay averages 4.5 days. Causes of prolonged rehabilitation period are often associated with severe pain syndrome, dyspepsia and postoperative complications. The complications rate after LC is about 6% and has no tendency to decrease. The implementation of enhanced recovery after surgery (ERAS) programs may potentially reduce stress-associated complications and improve the quality of rehabilitation. A few retrospective studies examined their advantages and setbacks in the treatment of acute cholecystitis with encouraging results. The aim of this randomized control study is to evaluate the modified ERAS program for patients with acute cholecystitis.

ELIGIBILITY:
Inclusion Criteria:

* Grade I and II acute cholecystitis according to Tokyo Guidelines 2013 classification (TG13)
* ASA I and II.

Exclusion Criteria:

* Severe acute cholecystitis (Grade III on TG13);
* Patient's refusal to participate;
* The language barrier;
* Transfer to the intensive care unit after surgery;
* ASA class ≥ III;
* Conversion to open procedure;
* Biliary hypertension detected during preoperative examination or intraoperatively.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 189 (Actual)
Dates: Start 2017-01-31 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2019-01-30 (Actual)

PRIMARY OUTCOMES:
Postoperative length of stay (pLOS) | 30 days
  Time interval measured from the end of the surgery until the moment of discharge from the hospital, measured in days

SECONDARY OUTCOMES:
Complication rate | 30 days
  Number of patients who develop postoperative complications (surgical site infections, intraabdominal organ-specific infection, postoperative ileus) in relation to the total number of patients, measured in percentage
Readmission rate | 30 days
  Number of patients with readmission to the hospital after discharge in relation to the total number of patients, measured as a percentage
Postoperative pain | 24 hours
  Level of postoperative pain syndrome measured with a visual analog scale in centimeters
Shoulder pain incidence | 24 hours
  Quantity of patients who developed shoulder pain after surgery in relation to the total number of patients, measured as a percentage
Shoulder pain level | 24 hours
  Level of shoulder pain syndrome measured with a visual analog scale in centimeters

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Sazhin, Prof., Study Chair — Pirogov Russian National Research Medical University
Locations (1):
- Taras Nechay, Moscow, Russia